CLINICAL TRIAL: NCT01977989
Title: Randomized Control Trial of Vancomycin Powder Following Posterior Instrumented Spinal Surgery for Trauma
Brief Title: Vancomycin in Spine Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Tennessee (Other)
Collaborators: Semmes-Murphey Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 13-02478-FB
Record Dates: First submitted 2013-10-31; First posted 2013-11-07 (Estimated); Last update posted 2013-11-07 (Estimated); Status verified 2013-10

CONDITIONS: Wound Infection
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No Vancomycin Powder (No Intervention): Patients who only receive IV Vancomycion prior to surgery. No Vancomycin powder is administered.
- Vancomycin Powder (Active Comparator): Patients who receive Vancomycin powder in the surgical site following surgery.
  Interventions: Drug: Vancomycin Powder

INTERVENTIONS:
Drug: Vancomycin Powder — For surgeries involving 3 contiguous spinal segments or less, 500mg of vancomycin will be applied topically. For surgeries involving more than 3 contiguous spinal segments, 1gm of vancomycin will be applied topically to the surgical site.
  Arms: Vancomycin Powder

SUMMARY:
The purpose of this study is to study how well using a powdered form of the antibiotic, vancomycin, inside the surgery wound prevents infection in patients undergoing instrumented spinal surgery for traumatic injury to the back.

Vancomycin is approved by the United States Food and Drug Administration (FDA) for treating certain kinds of bacteria. It is also used to prevent infections of the surgery site.

This will be a study in which the experimental treatment is compared to a standard (control) treatment. It will be prospective in nature, meaning that it will follow patients forward in time, and it will consist of a randomization process to determine who will receive the experimental treatment versus the standard (control) treatment.

The study will take place at Regional Medical Center (The MED). 140 subjects will be participating in this study.

The investigators hypothesize that the topical use of powder vancomycin will decrease the rate of surgical site infection.

DETAILED DESCRIPTION:
1. Purpose: The purpose of this study is to examine the efficacy of prophylactic, locally applied vancomycin powder against surgical site infection in patients undergoing posterior instrumented spinal surgery for traumatic injury.
2. Rationale: Surgical site infection (SSI) is a morbid complication with high cost in management of surgical spine patients. In this era of healthcare reforms, adjuvant therapies that not only improve quality, but also decrease cost, are considered of highest value. Despite the use of prophylactic systemic antibiotics and improved surgical technique, surgical site infections remain a serious perioperative concern. In comparison to systemic antibiotics, local delivery of antibiotics is attractive because high concentrations are achieved directly at these sites and systemic toxicity is limited.

   Prior investigations have primarily focused on the treatment of infected wounds with local antibiotics. Only a few studies have analyzed prophylactic use of local antibiotics during spine surgery. To date, there are no prospective, randomized studies on the prophylactic use of local antibiotics. The investigators will introduce local vancomycin powder into their practice of instrumented posterior spinal fusion for traumatic spine injury and determine efficacy in preventing postoperative infections.
3. Study Population: The study will consist of adult patients undergoing posterior, instrumented spine surgery for traumatic injury.
4. Research Design: This will be a prospective, randomized, controlled trial. The study will primarily be carried out through the University of Tennessee Health Science Center with all spinal surgery taking place at the Regional Medical Center at Memphis. Once patients with traumatic spine injury have been deemed eligible through several other criteria described later in the application, they will be placed into one of two randomized groups:

1) The control group will consist of patients who are administered systemic prophylactic antibiotic only.

2) The treatment group will consist of patients who are administered systemic prophylactic antibiotic along with vancomycin powder within the surgical site.

5. Study/Project Procedures: Patients who meet the entry criteria and agree to participate in the trial will be randomized to receive intraoperative vancomycin powder within the surgical wound or not. In all patients, vancomycin 1g and cefazolin 2g IV will be given within 60min of skin incision. If an allergy to cefazolin exists, 900mg of clindamycin IV will be used in its place. Cefazolin 1g IV will be given q6hr during surgery and continued q8hr post surgery for 24hrs, regardless of whether a surgical drain is in place. One to three liters of normal saline will be used for irrigation purposes during surgical procedure. Prior to wound closure, vancomycin powder will be topically applied both above (50% of dose) and below (50% of dose) the deep muscular fascia in patients participating in the treatment arm of the study. For surgeries involving 3 contiguous spinal segments or less, 500mg of vancomycin (1/2 vial) will be applied. For surgeries involving greater than 3 contiguous spinal segments, 1gm will be applied.

6. Outcome Measures: All patients will be followed on an inpatient or outpatient basis (as applicable) for a period of 12 months post-operatively. Residents, attendings and study coordinators will perform data collection. All patients with suspected wound infection will undergo MRI with contrast for verification, unless there is gross evidence of infection (ex. purulent drainage from the incision, erythema and swelling). A CT scan with contrast will be obtained in those patients who are unable to undergo MRI for various reasons (pacemaker, metallic foreign bodies, fresh vascular stents, etc.). All wound data will be collected and recorded in specific data forms at each clinical encounter.

ELIGIBILITY:
Inclusion Criteria:

* Hemodynamically stable
* 18 years of age or older
* Undergoing spinal fusion for traumatic cervical, thoracic, or lumbar injury

Exclusion Criteria:

* Septic patient
* Open or penetrating spinal injury
* Active infection
* Active cancer
* Known allergy to vancomycin
* Previous surgery in surgical site
* History of radiation therapy at surgical site
* Immunosuppressed (disease or drug-induced)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Surgical Site Infection | 12 Months
  All patients with suspected wound infection will undergo MRI with contrast for verification, unless there is gross evidence of infection. A CT scan with contrast will be obtained in those patients who are unable to undergo MRI for various reasons.

CONTACTS AND LOCATIONS:
Locations (1):
- Regional Medical Center (The MED), Memphis, Tennessee, United States

REFERENCES:
- [Background] Perencevich EN, Sands KE, Cosgrove SE, Guadagnoli E, Meara E, Platt R. Health and economic impact of surgical site infections diagnosed after hospital discharge. Emerg Infect Dis. 2003 Feb;9(2):196-203. doi: 10.3201/eid0902.020232. PMID 12603990
- [Background] Bibbo C, Patel DV. The effect of demineralized bone matrix-calcium sulfate with vancomycin on calcaneal fracture healing and infection rates: a prospective study. Foot Ankle Int. 2006 Jul;27(7):487-93. doi: 10.1177/107110070602700702. PMID 16842714
- [Background] Branstetter JG, Jackson SR, Haggard WO, Richelsoph KC, Wenke JC. Locally-administered antibiotics in wounds in a limb. J Bone Joint Surg Br. 2009 Aug;91(8):1106-9. doi: 10.1302/0301-620X.91B8.22216. PMID 19651846
- [Background] Buchholz HW, Engelbrecht H. [Depot effects of various antibiotics mixed with Palacos resins]. Chirurg. 1970 Nov;41(11):511-5. No abstract available. German. PMID 5487941
- [Background] Calderone RR, Garland DE, Capen DA, Oster H. Cost of medical care for postoperative spinal infections. Orthop Clin North Am. 1996 Jan;27(1):171-82. PMID 8539047
- [Background] Burdon DW. Principles of antimicrobial prophylaxis. World J Surg. 1982 May;6(3):262-7. doi: 10.1007/BF01653540. No abstract available. PMID 7113232
- [Background] Cavanaugh DL, Berry J, Yarboro SR, Dahners LE. Better prophylaxis against surgical site infection with local as well as systemic antibiotics. An in vivo study. J Bone Joint Surg Am. 2009 Aug;91(8):1907-12. doi: 10.2106/JBJS.G.01237. PMID 19651948
- [Background] Dahners LE, Funderburk CH. Gentamicin-loaded plaster of Paris as a treatment of experimental osteomyelitis in rabbits. Clin Orthop Relat Res. 1987 Jun;(219):278-82. PMID 3581579
- [Background] Edin ML, Miclau T, Lester GE, Lindsey RW, Dahners LE. Effect of cefazolin and vancomycin on osteoblasts in vitro. Clin Orthop Relat Res. 1996 Dec;(333):245-51. PMID 8981903
- [Background] Gitelis S, Brebach GT. The treatment of chronic osteomyelitis with a biodegradable antibiotic-impregnated implant. J Orthop Surg (Hong Kong). 2002 Jun;10(1):53-60. doi: 10.1177/230949900201000110. PMID 12401922
- [Background] Glassman SD, Dimar JR, Puno RM, Johnson JR. Salvage of instrumental lumbar fusions complicated by surgical wound infection. Spine (Phila Pa 1976). 1996 Sep 15;21(18):2163-9. doi: 10.1097/00007632-199609150-00021. PMID 8893444
- [Background] Gold HS, Moellering RC Jr. Antimicrobial-drug resistance. N Engl J Med. 1996 Nov 7;335(19):1445-53. doi: 10.1056/NEJM199611073351907. No abstract available. PMID 8875923
- [Background] Isefuku S, Joyner CJ, Simpson AH. Gentamicin may have an adverse effect on osteogenesis. J Orthop Trauma. 2003 Mar;17(3):212-6. doi: 10.1097/00005131-200303000-00010. PMID 12621263
- [Background] Isefuku S, Joyner CJ, Simpson AH. Toxic effect of rifampicin on human osteoblast-like cells. J Orthop Res. 2001 Sep;19(5):950-4. doi: 10.1016/S0736-0266(01)00022-5. PMID 11562146
- [Background] Klemm KW. Antibiotic bead chains. Clin Orthop Relat Res. 1993 Oct;(295):63-76. PMID 8403672
- [Background] Levi AD, Dickman CA, Sonntag VK. Management of postoperative infections after spinal instrumentation. J Neurosurg. 1997 Jun;86(6):975-80. doi: 10.3171/jns.1997.86.6.0975. PMID 9171176
- [Background] Martin C, Viviand X, Potie F. Local antibiotic prophylaxis in surgery. Infect Control Hosp Epidemiol. 1996 Aug;17(8):539-44. doi: 10.1086/647366. PMID 8875300
- [Background] Hanssen AD. Local antibiotic delivery vehicles in the treatment of musculoskeletal infection. Clin Orthop Relat Res. 2005 Aug;(437):91-6. doi: 10.1097/01.blo.0000175713.30506.77. PMID 16056032
- [Background] Holtom PD, Pavkovic SA, Bravos PD, Patzakis MJ, Shepherd LE, Frenkel B. Inhibitory effects of the quinolone antibiotics trovafloxacin, ciprofloxacin, and levofloxacin on osteoblastic cells in vitro. J Orthop Res. 2000 Sep;18(5):721-7. doi: 10.1002/jor.1100180507. PMID 11117292
- [Background] Hou T, Xu J, Li Q, Feng J, Zen L. In vitro evaluation of a fibrin gel antibiotic delivery system containing mesenchymal stem cells and vancomycin alginate beads for treating bone infections and facilitating bone formation. Tissue Eng Part A. 2008 Jul;14(7):1173-82. doi: 10.1089/ten.tea.2007.0159. PMID 18593356
- [Background] Sweet FA, Roh M, Sliva C. Intrawound application of vancomycin for prophylaxis in instrumented thoracolumbar fusions: efficacy, drug levels, and patient outcomes. Spine (Phila Pa 1976). 2011 Nov 15;36(24):2084-8. doi: 10.1097/BRS.0b013e3181ff2cb1. PMID 21304438
- [Background] O'Neill KR, Smith JG, Abtahi AM, Archer KR, Spengler DM, McGirt MJ, Devin CJ. Reduced surgical site infections in patients undergoing posterior spinal stabilization of traumatic injuries using vancomycin powder. Spine J. 2011 Jul;11(7):641-6. doi: 10.1016/j.spinee.2011.04.025. Epub 2011 May 19. PMID 21600853
- [Background] Kirkland KB, Briggs JP, Trivette SL, Wilkinson WE, Sexton DJ. The impact of surgical-site infections in the 1990s: attributable mortality, excess length of hospitalization, and extra costs. Infect Control Hosp Epidemiol. 1999 Nov;20(11):725-30. doi: 10.1086/501572. PMID 10580621